CLINICAL TRIAL: NCT06478537
Title: Thrombopoietin Receptor Agonist (TPO-RA) Treatment on Immune Tolerance Induction of ITP Patients With Sustained Platelet Recovery After Treatment Termination
Brief Title: TPO-RA Treatment on Immune Tolerance Induction of ITP Patients With Sustained Platelet Recovery After Treatment Termination
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Tienan Zhu, Director, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-24PJ1123
Record Dates: First submitted 2024-06-13; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; thrombopoietin receptor agonist (TPO-RA); hetrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — hetrombopag; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hetrombopag treatment (Experimental)
  Interventions: Drug: Hetrombopag Olamine; Drug: Aspirin

INTERVENTIONS:
Drug: Hetrombopag Olamine — Treatment period: 24-week Hetrombopag (2.5mg/d~7.5mg/d) treatment.
  * Two consecutive visits with PLT>600 × 10^9/L: daily dose reduction of 2.5mg; If the lowest dose has been used, extend the dosing interval.
  * Two consecutive visits with PLT<300 × 10^9/L: increase the daily dose by 2.5mg until the maximum dose is reached.
  * Two consecutive visits with PLT<50 × 10^9/L: increase the daily dose by 2.5mg until the maximum dose is reached; If PLT is still<50 × 10^9/L with7.5mg/d × 28d, the patient will be withdrawn.
  Drug discontinuation period：8-week Hetrombopag (2.5mg/d~7.5mg/d) reduction. Hetrombopag reduces by 2.5mg every 2 weeks, and after reducing to the minimum dose of 2.5mg/d x 2 weeks, it is changed to 2.5mg once every other day (Qod) treatment, with a maximum reduction time of 8 weeks. If the PLT during two consecutive visits is less than 30 × 10^9/L, the patient will be withdrawn.
  Other Names: Hetrombopag
Drug: Aspirin — Aspirin 100mg, qd

SUMMARY:
The aim of this study was to observe whether maintaining a high level of platelet count after TPO-RA in patients with primary immune thrombocytopenia (ITP) can induce immune tolerance, develop immune balance in ITP patients, and enable patients to achieve a sustained response (SRoT) after TPO-RA discontinuation.

DETAILED DESCRIPTION:
In this study, ITP patients who has reached complete response (PLT ≥100 x 10^9/L）after thrombopoietin receptor agonist (TPO-RA) therapy do not rush to reduce the drug dose, so that a higher level of platelet count can be maintained for a period of time.

The treatment goal is to maintain the patient's platelet count at 300-600 × 10^9/L, and adjust the dosage of hetrombopag (2.5mg/d~7.5mg/d) based on the patient's platelet count. After 24-week TPO-RA treatment, all patients with a platelet count of ≥ 50 × 10^9/L after two consecutive visits will enter an 8-week reduction period. All patients who successfully discontinued the drug and maintained their platelet count at ≥30×109/L entered the efficacy and safety follow-up period.

The aim is to investigate whether this strategy could lead to the development or achievement of immune tolerance, achieving sustained response off treatment (SROT) (PLT≥50×109/L, no other ITP-specific medications, no bleeding) after TPO-RA discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of gender;
2. Patients with newly diagnosed or persistent primary ITP who have shown inadequate response or relapse following first-line corticosteroid treatment with or without IVIg;
3. Complete response (PLT > 100 × 10^9/L) achieved after hetrombopag treatment at doses of 2.5mg-7.5mg per day;
4. Volunteer to participate in clinical research and sign an informed consent form, willing to follow and capable of completing all trial procedures.

Exclusion Criteria:

1. Age>50 years old;
2. Those who are contraindicated to taking aspirin;
3. Previous arterial or venous thrombosis history (including coronary atherosclerotic heart disease, ischemic stroke, deep vein thrombosis or pulmonary embolism, etc.) or clinical symptoms and medical history indicate thrombophilia;
4. Risk factors of cardiovascular diseases such as hypertension, diabetes and hyperlipidemia;
5. Heart disease occurring within the first 3 months of screening, including congestive heart failure classified as III/IV by the New York Heart Association (NHYA), arrhythmias or myocardial infarction requiring medication, or arrhythmias known to increase the risk of thrombotic events (such as atrial fibrillation), or prolonged QT interval (QTc) after subject correction (QTc>450 milliseconds, or QTc>480 milliseconds in subjects with bundle branch block)
6. Patients currently undergoing anticoagulant therapy or antiplatelet therapy;
7. Female patients receiving estrogen replacement therapy or oral contraceptives;
8. Patients with past or current malignant tumors;
9. Secondary thrombocytopenia, such as myelodysplastic syndrome, immune disorders such as systemic lupus erythematosus, early aplastic anemia, atypical aplastic anemia, antiphospholipid syndrome, thrombotic thrombocytopenic purpura, and other causes of thrombocytopenia;
10. The results of bone marrow biopsy during the screening period indicate that the bone marrow fibrosis MF is ≥ 2 (Thieleja 2005, the European expert consensus bone marrow fibrosis scoring standard), or that bone marrow biopsy suggests the presence of other primary diseases that can cause thrombocytopenia besides ITP;
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are three times higher than the upper limit of normal values, total bilirubin is three times higher than the upper limit of normal values, and blood creatinine is 1.5 times higher than the upper limit of normal values;
12. Have a history of liver cirrhosis or portal hypertension;
13. Uncontrollable infections;
14. Hepatitis B surface antigen positive or previous history of hepatitis B, and in the past 3 months, accompanied by HBV-DNA ≥ 2000IU/ML; those with positive hepatitis C antibody, HCV-RNA positive in the past 3 months;
15. Individuals who test positive for antibodies against human immunodeficiency virus or specific antibodies against Treponema pallidum;
16. Individuals who are known to be allergic to the drug itself or its excipients;
17. Breastfeeding or pregnant women or female patients planning to conceive during the study period; 18）Other situations determined by the researcher as unsuitable for participation in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Sustained response off treatment (SROT) | 3 year
  The percentage of participants with successful discontinuation of TPO-RAs after tapering and discontinuation

SECONDARY OUTCOMES:
Quality of life (QoL) | 3 year
  The degree to which an individual is healthy, comfortable, and able to participate in or enjoy life events according to the MOS 36-item short-form health survey (SF-36) at week1, week24 and week56 (±5 d).
Duration of Complete response (DCR) | 3 year
  The time from the first assessment of complete resonse (platelet count ≥ 100 × 10^9/L, without bleeding) until the date of the first occurrence of progression, or until the date of death.t
Duration of Response (DoR) | 3 year
  The time from the first assessment of response (platelet count ≥ 50 × 10^9/L) until the date of the first occurrence of progression, or until the date of death.
Adverse events | 3 years
  The incidence and severity of thromboembolism, as well as other commonly used indicators such as abnormal clinical symptoms and vital signs, abnormalities observed in laboratory tests, are recorded.Toxicity will be graded according to NCI-CTC AE 5.0.
Bleeding events | 3 years
  Bleeding events occurring in patients due to ITP

CONTACTS AND LOCATIONS:
Overall Officials: Tienan Zhu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China